CLINICAL TRIAL: NCT04432532
Title: Neuroendocrine and Adrenal Tumors: Biochemical, Histopathologic and Genetic Studies
Brief Title: Neuroendocrine and Adrenal Tumors
Acronym: NETAT
Status: Withdrawn | Type: Observational
Why Stopped: Change in research direction
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Heather Wachtel, MD, Assistant Professor of Surgery, University of Pennsylvania
Other Study IDs: 832475
Record Dates: First submitted 2020-03-09; First posted 2020-06-16 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors; Adrenal Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor specimens, blood and/or saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuroendocrine Tumor
  Interventions: Other: No intervention
- Adrenal Tumor
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There are no interventions

SUMMARY:
This is a prospective study of rare neuroendocrine and adrenal tumors. Subjects will be enrolled via informed consent, and blood and/or saliva and tissue will be collected. This is designed to work in conjunction with IRB#831990 which is a retrospective protocol. The University of Pennsylvania will be a contributing site with the University of Michigan as the coordinating site for the A5 alliance, a multi-institutional collaborative designed to study neuroendocrine and adrenal tumors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with neuroendocrine and/or an adrenal tumor

Exclusion Criteria:

* pregnant women
* prisoners
* people under the age of 18

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and seeking treatment for neuroendocrine tumors or adrenal tumors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years

SECONDARY OUTCOMES:
Tumor Recurrence | 10 years
  We want to record recurrences in our patient population

IPD SHARING:
Plan to Share IPD: Yes